CLINICAL TRIAL: NCT05157958
Title: Double Blind, Randomized, Phase II Clinical Study to Evaluate Safety and Efficacy of ALLO-ASC-SHEET Versus Vehicle Control in Dystrophic Epidermolysis Bullosa (DEB) Patients
Brief Title: Study to Evaluate Safety and Efficacy of ALLO-ASC-SHEET in Subjects With Dystrophic Epidermolysis Bullosa
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Anterogen Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ALLO-ASC-DEB-201
Record Dates: First submitted 2021-12-02; First posted 2021-12-15 (Actual); Last update posted 2024-04-22 (Actual); Status verified 2024-04

CONDITIONS: Dystrophic Epidermolysis Bullosa
MeSH Terms: conditions — Epidermolysis Bullosa Dystrophica

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ALLO-ASC-SHEET (Experimental): Allogeneic mesenchymal stem cells
  Dressing for Dystrophic Epidermolysis Bullosa wound
  Interventions: Biological: ALLO-ASC-SHEET
- Conventional Therapy (Active Comparator): Hydrogel Sheet
  Matching control
  Interventions: Other: Vehicle Control

INTERVENTIONS:
Biological: ALLO-ASC-SHEET — Weekly administration
  Arms: ALLO-ASC-SHEET
Other: Vehicle Control — Weekly administration
  Arms: Conventional Therapy

SUMMARY:
After confirming eligibility, a single subject with four selected target lesions will receive both ALLO-ASC-SHEET and Vehicle control, three target lesions for ALLO-ASC-SHEET and the other target for Vehicle control, and which lesion to apply which IP treatment will be determined randomly at the time of enrollment using pre-designed block randomization scheme.

DETAILED DESCRIPTION:
Primary efficacy endpoint will be assessed during and after 12th IP applications.

ELIGIBILITY:
Key Inclusion Criteria:

1. Subject diagnosed as dystrophic epidermolysis bullosa confirmed by clinical criteria and one of the following:

   1. Immunostaining test: patients who have reduced or no type 7 collagen in staining degree of immunofluorescence. Other antigens (laminin-332, type 17 collagen, plectin, integrin α6β4, type 5 and type 14 keratin, etc.) are normal in immune-staining.
   2. COL7A1 mutational analysis: confirmation of COL7A1 genetic mutation.
2. Subject with skin ulcer lesions of dystrophic epidermolysis bullosa meet the following criteria, on the screening start day (Visit 1) and treatment start day (enrollment day) (Visit 3):

   1. Subject has two skin ulcer lesions judged as comparable to compare the safety and efficacy by investigator during screening period and prior to the IP application (enrollment day).
   2. Two skin ulcer lesions meeting criteria stated in 2a) should be sized 5-20 cm2 (inclusive)
3. Subject who has two comparable target skin ulcer lesions, and each lesions with a change of size equal to or less than ±50% at treatment day (Visit 3) compared to that of screening day (Visit 1)
4. Subject who has no clinical evidence of infection related signs/symptoms, or visible necrosis in the target skin ulcer area (area including ulcer lesion and surrounding area where the IP is to be applied).

Key Exclusion Criteria:

1. Subject who requires antibiotics due to bacterial infection on skin of the target skin ulcer area (area including ulcer lesion and surrounding area where the IP is to be applied).
2. Female subjects: pregnant woman (indicated by serum hCG test result at screening), breast-feeding patient, all sexually active patient, with child bearing potential in case of female*, who is not willing to contracept** during the clinical trial.

Ages: 4 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-10-01 (Estimated); Study Completion 2026-04-28 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | First application to week 37
  Incidence, severity, relationship of adverse event

SECONDARY OUTCOMES:
Proportion of complete wound closure | First application to week 17
  Proportion of subject with target skin ulcer area meeting the definition of wound closure during and at the completion of 12 weeks treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of Miami Dermatology Clinical Trials Unit, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: No